CLINICAL TRIAL: NCT06874491
Title: Effects of Two Different Distraction Methods on Fear and Anxiety Levels in Preschool Children Receiving Inhalation Treatment
Brief Title: Inhalation Treatment Distraction in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/136
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-03

CONDITIONS: Fear Anxiety

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Moving and 3D Book Group (Experimental): After the data collector is taken to the environment where the child will receive inhalation treatment, the child and the parent will be introduced and the purpose of the study will be explained and the scales will be filled. During the inhaler treatment, the researcher will ensure that the child spends time with a moving and 3D book that will be specially designed and suitable for inhalation treatment. After the treatment is completed, the child's reactions will be evaluated and the scales will be filled again. Filling out the forms will take approximately 5-10 minutes.
  Interventions: Behavioral: Moving and 3D Book
- Hand Puppet Group (Experimental): After the data collector is taken to the environment where the child will receive inhalation treatment, the child and parent will be introduced and the purpose of the study will be explained and the scales will be filled. During the inhaler treatment, the researcher will ensure that the child spends time with a hand puppet that will be specially designed and suitable for inhalation treatment. After the treatment is completed, the child's reactions will be evaluated and the scales will be filled again. Filling out the forms will take approximately 5-10 minutes.
  Interventions: Behavioral: Hand Puppet
- Control Group (No Intervention): The data collector will be taken to the environment where the child will receive inhalation treatment and the routine procedures will be continued. Then, the child and the parent will be introduced and the purpose of the study will be explained and the scales will be filled. After the treatment is completed, the child's reactions will be evaluated and the scales will be filled again. Filling out the forms will take approximately 5-10 minutes.

INTERVENTIONS:
Behavioral: Moving and 3D Book — After the data collector is taken to the environment where the child will receive inhalation treatment, the child and the parent will be introduced and the purpose of the study will be explained and the scales will be filled out. During the inhaler treatment, the child will spend time with a moving and 3D book that will be specially designed for inhalation treatment. After the treatment is completed, the child's reactions will be evaluated and the scales will be filled out again. Filling out the forms will take an average of 5-10 minutes.
  Arms: Moving and 3D Book Group
Behavioral: Hand Puppet — After the data collector is taken to the environment where the child will receive inhalation treatment, the child and the parent will be introduced and the purpose of the study will be explained and the scales will be filled out. During the inhaler treatment, the child will spend time with a hand puppet that will be specially designed for inhalation treatment by the researcher. After the treatment is completed.
  Arms: Hand Puppet Group

SUMMARY:
The aim of the project is to examine the effects of two different distraction methods used in preschool children receiving inhalation therapy on fear and anxiety levels. Children are exposed to various hospital procedures throughout their lives. These procedures cause children to experience fear, pain and anxiety. One of these procedures is inhalation therapy. When children wear the face masks required for inhalation, they experience intense fear and anxiety. Non-pharmacological techniques are used for the effective management of this fear and anxiety. Among these techniques, distraction is the easy-to-apply. When applying distraction techniques, the child's developmental period, age group and interest should be taken into consideration. The project is a randomized controlled trial. The universe of the study will consist of children between the ages of 4-6 who received inhalation therapy for the first time in the pediatric emergency department of Erzincan Mengücek Gazi Education and Research Hospital between September 2025 and September 2026. In collecting the research data, "Questionnaire Form", "Child Fear Scale" and "Child Anxiety Scale-State" will be used.

The two different methods to be used will be designed to attract the attention and interest of the age groups of the children to be included in the research. In this way, it is thought that the child will focus his/her attention and curiosity on the two different methods to be used and the level of fear and anxiety will be affected during the inhalation treatment. This will increase the child's compliance and cooperation with the treatment and will encourage the child.

When the international and national literature was scanned, no study was found that investigated the effects of the two different distraction methods covered in the research during inhalation treatment. With the two different distraction methods to be used, inhalation treatment, which is a source of fear and anxiety for children, will become fun.

DETAILED DESCRIPTION:
Children are exposed to various hospital procedures throughout their lives. These procedures cause children to experience fear, pain and anxiety. One of these procedures is inhalation therapy. When children wear the face masks required for inhalation, they experience intense fear and anxiety. Non-pharmacological techniques are used for the effective management of this fear and anxiety. Among these techniques, distraction is the easy-to-apply. When applying distraction techniques, the child's developmental period, age group and interest should be taken into consideration. The project is a randomized controlled trial. The universe of the study will consist of children between the ages of 4-6 who received inhalation therapy for the first time in the pediatric emergency department of Erzincan Mengücek Gazi Education and Research Hospital between September 2025 and September 2026. In collecting the research data, "Questionnaire Form", "Child Fear Scale" and "Child Anxiety Scale-State" will be used.

Movable and 3D book: Movable and 3D book that will be suitable and specially designed for inhalation therapy will be used. The book will include materials that children frequently encounter in inhalation therapy (mask, nebulizer, drug models used for treatment, a model of the nurse administering the treatment, and a model of the environment where inhalation therapy is performed). The book is aimed to attract children's attention by being made in an animated and three-dimensional form. The prepared book is presented to the opinions of experts in the field of child health and improvements will be made in line with the feedback. The final version of the book, which is specially designed and suitable for inhalation therapy, will be converted into two different formats and made ready for use in research. The aim of preparing it in two formats is to increase the child's interest in the book by giving him the right to choose. It is thought that this innovative book will have significant effects on children's fear and anxiety levels.

Hand Puppet: A hand puppet that is specially designed for inhalation therapy will be used. Hand puppets that aim to make inhalation therapy fun will be prepared (by playing with children the situations of different characters receiving inhalation therapy in the form of a game). The hand puppets that will be designed with the researcher, preschool teacher and child development specialist who receive play therapy will be prepared in a hypoallergenic form. In order to provide children with the right to choose, different forms will be prepared and children's ideas will be given importance. It is thought that the hand puppet that is specially designed for inhalation therapy will have significant effects on children's fear and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* -Being between 4-6 years old
* Not having a developmental disability
* Not having a history of sedative, analgesic or narcotic substance use within 24 hours before application
* Receiving inhalation therapy for the first time
* Not having a chronic disease
* Children who are accompanied by their mother or father during the procedure will be included in the study.

Exclusion Criteria:

* Being under 4 years old or over 6 years old
* having a chronic disease

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Child Fear Scale | 1 YEAR
  The Child Fear Scale was developed by McMurty and colleagues in 2011 to measure fear in children undergoing painful medical procedures. The Turkish validity and reliability of the scale was performed by Özalp Gerçeker and colleagues in 2018. The Child Fear Scale is a 0-4 scale showing five faces ranging from a neutral expression (0 = no anxiety at all) to the feared face (4 = severe anxiety).
Child Anxiety Scale-State | 1 YEAR
  The scale, developed by Ersig and his colleagues in 2013, was validated in Turkish by Özalp Gerçeker and his colleagues in 2018. The "Children's Anxiety Scale-State, which resembles a thermometer with horizontal lines, is scored from 0 to 10. It is a scale developed for children aged 4 to 10. When the scale is introduced to the child, it is said that there is no anxiety, that anxiety increases as it goes up, and that the anxiety level is very high at the top. The child is then asked to draw a line in the section that shows how anxious or nervous he is.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.